CLINICAL TRIAL: NCT04626752
Title: An Open, Uncontrolled, Multicenter Clinical Trial to Explore the Safety, Efficacy, and Remission Phase of Chimeric Antigen Receptor T Cell (CAR-T) in the Treatment of Relapsed Refractory (R/R) Multiple Myeloma (MM)
Brief Title: CAR-T Cells in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR-T for Multiple myeloma
Record Dates: First submitted 2020-11-06; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — fludarabine; Influenza Vaccines; Cyclophosphamide; Cholestanetriol 26-Monooxygenase

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- volunteers (Experimental): The patient voluntarily signs the informed consent, and the patient meets the entry criteria to diagnose patients with Relapsed Refractory (R/R) Multiple Myeloma (MM)
  Interventions: Drug: BCMA CAR-T; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: BCMA CAR-T — Volunteers will be treated with BCMA CAR-T cells
  Other Names: senl_BCMA
Drug: Fludarabine — 25mg/㎡ for D-4、D-3 and D-2
  Other Names: flu
Drug: Cyclophosphamide — 500mg/㎡ for D-3 and D-2
  Other Names: ctx

SUMMARY:
This study is aimed to evaluate the safety, feasibility and efficacy of CAR-T cell therapy in the treatment of relapsed or refractory multiple myeloma

DETAILED DESCRIPTION:
This is a study to evaluate the safety, feasibility and efficacy of CAR-T cell therapy in the treatment of relapsed or refractory multiple myeloma.

The Main research objectives:

To evaluate the safety and efficacy of CAR-T cell therapy in patients with relapsed or refractory multiple myeloma.

The Secondary research objectives:

To evaluate the safety and efficacy of CAR-T cell therapy in patients with relapsed or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily participated in the study and signed the informed consent form by themselves or their legal guardian;
2. According to the international standard for multiple myeloma (IMWG 2014);
3. Diagnosed as relapsed or refractory multiple myeloma. Relapsed and refractory were defined as follow.

   Relapsed: patients had received for at least 3 drugs with different mechanisms of action (including protease inhibitors and immunomodulators) and disease progression within 60 days of the most recent treatment. Refractory was defined as: disease progression occurred during the recent treatment, or disease progression occurred within 60 days after treatment;
4. The expression of BCMA in myeloma cells was reported as positive by flow cytometry or immunohistochemistry;
5. No antibody drug was administered within last 2 weeks before cell therapy;
6. ECOG Scores: 0~1
7. Echocardiography showed normal diastolic function, left ventricular ejection fraction (LVEF) ≥ 50%, no serious arrhythmia;
8. The subjects had no pulmonary infection, normal pulmonary function, and indoor air oxygen saturation ≥92%;
9. There was no contraindication for peripheral blood sampling;
10. The estimated survival time was more than 12 weeks;
11. The urine pregnancy test of female subjects of childbearing age should be negative and not in lactation; the female or male subjects of childbearing age should take effective contraceptive measures during the whole research process.

Exclusion Criteria:

1. Have a history of allergy to any component of cell products;
2. There are clinically significant cardiovascular diseases, such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or any grade 3 (moderate) or grade 4 (severe) heart disease with cardiac function (according to the functional classification method of the New York Heart AssociationNYHA) with a history of myocardial infarction, angioplasty or stent implantation, unstable angina or other clinically significant heart disease within 12 months before admission;
3. who has suffered from brain injury, consciousness disorder, epilepsy, more serious cerebral ischemia or cerebral hemorrhage disease;
4. Patients who need urgent treatment due to tumor progression or spinal cord compression;
5. The investigator determines that there are serious complications or diseases that will increase the risk of the subject or affect the study, including but not limited to, for example, cirrhosis, recent major trauma, etc;
6. After allogeneic hematopoietic stem cell transplantation;
7. Patients with autoimmune diseases, immunodeficiency or other diseases requiring immunosuppressive（excluding glucocorticoid）therapy;
8. There was uncontrolled active infection;
9. There were live vaccinations within 4 weeks before admission;
10. Active hepatitis (positive for HBVDNA or HCVRNA), syphilis and other acquired and congenital immunodeficiency diseases, including but not limited to those with HIV infection;
11. Subjects had a history of alcohol, drug or mental illness;
12. The researchers believe that there are other conditions that subjects are not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Severe/Adverse Events as a Measure of Safety | 28 days
  Number of Participants with Severe/Adverse Events as a Measure of Safety
CAR-T Cell expansion level | 24 months
  Copies numbers of CAR in peripheral blood(PB) and/or bone marrow(BM)

SECONDARY OUTCOMES:
Objective response rate of complete remission and partial remission | 24 months
  Objective response rate of complete remission and partial remission
Overall survival time | 24 months
  Overall survival time

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Luo, PhD&MD, Principal Investigator — The Second Hospital of Hebei Medical University
Locations (1):
- the Second Hospital of HeBei Medical University (HBMU), Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No